CLINICAL TRIAL: NCT03320161
Title: A Patient Consensus for the Research in Supportive Care in French Cancer Care Centers: the CyPRES Project
Acronym: CyPRES
Status: Completed | Type: Observational
Sponsor: UNICANCER (Other)
Collaborators: Ligue contre le cancer, France (Other); French National Platform Quality of Life and Cancer (Unknown); Association Francophone des Soins Oncologiques de Support (Unknown)
Responsible Party: Sponsor
Other Study IDs: UC-0106/1707
Record Dates: First submitted 2017-10-20; First posted 2017-10-25 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Cancer Patients
Keywords: Supportive care; Cancer; Health-related quality of life; Consensus; Participative approach; Patient involvement; DELPHI method
MeSH Terms: conditions — Neoplasms; Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In oncology a number of supportive care therapies are proposed to patients. This study will identify the different therapies and prioritize these therapies from the patients' perspectives. This study will provide a framework for optimizing supportive care strategies and identifying those therapies that need to be validated by clinical trials.

DETAILED DESCRIPTION:
In oncology, supportive care should be used along with curative treatment or palliative care in order to improve patients' health-related quality of life, overall survival and to better support treatment side effects as well as the disease evolution. Unfortunately, they are not widely used in clinical practice.

A direct assessment of the needs perceived unmet by patients could allow to assess the magnitude of expectations to better target treatments as example. A prospective assessment of the expectations and needs of the patients is thus essential. This would also allow help to highlight the convergence between supportive care proposed and used and those expected by patients. The first step to understanding how to optimize the use of resources and to improve the quality of care is to identify patient's expectations. Moreover, it is now well recognized that patients should play a key role in the research and that their active participation in research can increase the relevance of the research.

In this context, the CyPRES project aims to:

1. assess through national consensus the patients' expectations in terms of supportive care in order to help both clinicians and health care services;
2. prioritize them and to arrange resources according to priority needs identified;
3. identify supportive care for which no previous research (evidence-based medicine) has demonstrated their usefulness. A randomized clinical trial will thus be proposed;
4. Involve patients in the written, conduct and analyses, as well as communications of the randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* patients supported for cancer
* patients of ERI, Espaces Ligue (french cancer care centers) or patient associations
* patients aged at least 18 years old

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients of french cancer care centers (ERI, Espaces Ligue) or patients Associations will be asked to answer the two questionnaires
Sampling Method: Probability Sample
Enrollment: 604 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Supportive care listed and prioritized by patients | At inclusion visit
  Expectations and needs of the patients: completion of questionnaire N°1
Supportive care listed and prioritized by patients | 4 to 7 months after inclusion
  Prioritize supportive care therapies: completion of questionnaire N°2 Expectations and needs of the patients questionnaire n°2 completed

CONTACTS AND LOCATIONS:
Overall Officials: Amélie Anota, PhD, Principal Investigator — Mehodology and Quality of Life in Oncology unit, CHRU Besançon, France
Locations (58):
- France (56):
  - Ligue Nationale Contre le Cancer - Comité de la Somme, Amiens
  - ICO - Site Paul Papin, Angers
  - Ligue Nationale Contre le Cancer - Comité du Maine-et-Loire, Angers
  - Ligue Nationale Contre le Cancer - Comité de Charente, Angoulême
  - Ligue Nationale Contre le Cancer - Comité du Val d'Oise, Argenteuil
  - Ligue Nationale Contre le Cancer - Comité des Pyrénées Atlantiques, Bayonne
  - Ligue Nationale Contre le Cancer - Comité de l'Oise, Beauvais
  - Institut Bergonié, Bordeaux
  - Ligue Nationale Contre le Cancer - Comité du Finistère, Brest
  - Ligue Nationale Contre le Cancer - Comité de l'Essonne, Briis-sous-Forges
  - Ligue Nationale Contre le Cancer - Comité du Lot, Cahors
  - Ligue Nationale Contre le Cancer - Comité du Puy-de-Dôme, Chamalières
  - Pôle Santé Léonard de Vinci, Chambray-lès-Tours
  - Centre Jean Perrin, Clermont-Ferrand
  - Ligue Nationale Contre le Cancer - Comité du Val-de-Marne, Créteil
  - Ligue Nationale Contre le Cancer - Comité des Landes, Dax
  - Ligue Nationale Contre le Cancer - Comité des Alpes de Haute-Provence, Digne-les-Bains
  - Ligue Nationale Contre le Cancer - Comité de la Côte-d'Or, Dijon
  - Centre Georges François Leclerc, Dijon
  - Ligue Nationale Contre le Cancer - Comité des Vosges, Épinal
  - Hôpital du Bocage, Grenoble
  - Ligue Nationale Contre le Cancer - Comité de la Vendée, La Roche-sur-Yon
  - Ligue Nationale Contre le Cancer - Comité de Seine-Saint-Deniss, Le Bourget
  - Ligue Nationale Contre le Cancer - Comité de la Haute-Vienne, Limoges
  - Ligue Nationale Contre le Cancer - Comité du Rhône, Lyon
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Ligue Nationale Contre le Cancer - Comité de Moselle, Metz
  - CHRU Montpellier - Hôpital Saint Eloi, Montpellier
  - Ligue Nationale Contre le Cancer - Comité de l'Hérault, Montpellier
  - Hôpital Emile Muller, Mulhouse
  - CHU de Nantes - Hôpital Dieu, Nantes
  - Hôpital Privé du Confluent, Nantes
  - Centre Antoine Lacassagne, Nice
  - Ligue Nationale Contre le Cancer - Comité du Gard, Nîmes
  - ERI Territorial du Gard - Institut de Cancérologie du Gard, Nîmes
  - Ligue Nationale Contre le Cancer - Comité de Paris, Paris
  - Institut Curie, Paris
  - Ligue Nationale Contre le Cancer - Comité des Pyrénées Atlantiques, Pau
  - Pôle Régional de Cancérologie - CHU Poitiers, Poitiers
  - Ligue Nationale Contre le Cancer - Comité de l'Ardèche, Privas
  - Ligue Nationale Contre le Cancer - Comité de la Marne, Reims
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Ligue Nationale Contre le Cancer - Comité de Seine-Maritime, Rouen
  - Ligue Nationale Contre le Cancer - Comité des Côtes-d'Armor, Saint-Brieuc
  - Ligue Nationale Contre le Cancer - Comité de la Loire, Saint-Etienne
  - Institut de Cancérologie de l'Ouest - ICO - René Gauducheau, Saint-Herblain
  - Institut de Cancérologie de la Loire - Lucien Neuwirth, Saint-Priest-en-Jarez
  - Centre Paul Strauss, Strasbourg
  - Ligue Nationale Contre le Cancer - Comité des Hautes-Pyrénées, Tarbes
  - Polyclinique de l'Ormeau, Tarbes
  - Ligue Nationale Contre le Cancer - Comité de l'Aube, Troyes
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Ligue Nationale Contre le Cancer - Comité des Yvelines, Versailles
  - Institut Gustave Roussy, Villejuif
- Martinique (2):
  - Ligue Nationale Contre le Cancer - Comité de la martinique, Fort-de-France
  - Centre Hospitalier Universitaire de Martinique, Fort-de-France

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.